CLINICAL TRIAL: NCT03673891
Title: Evaluation of Fluid Infusion With LifeFlow for Patients With Suspected Septic Shock
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Srikar Adhikari, Associate Professor, University of Arizona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 188903474
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Sepsis; Volume Assessment
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): After obtaining the consent, the subject will have a bedside ultrasound performed by the study investigator after receiving 500 ml of intravenous fluid bolus. The images will be recorded on ultrasound machine hard drive for future review. If the bedside ultrasound findings determine that the subject is not fluid responsive, subjects will be excluded from the study. If the subject is determined to be fluid responsive, the above listed outcome measures will be collected. Ultrasound will be repeated after every 500 ml bolus if the patient continues to receive IV fluids which will be determined by the treating physician. Ultrasound measurements and other parameters listed above will be collected throughout the ED and hospital stay.
- LifeFlow group (Experimental): LifeFlow device will be used to administer intravenous fluids in this group. LifeFlow is a FDA approved device to administer IV fluids. Subject will have a bedside ultrasound performed by the study investigator after receiving 500 ml of intravenous fluid bolus. The images will be recorded on ultrasound machine hard drive for future review. If the bedside ultrasound findings determine that the subject is not fluid responsive, subjects will be excluded from the study. If the subject is determined to be fluid responsive, the above listed outcome measures will be collected. Ultrasound will be repeated after every 500 ml bolus if the patient continues to receive IV fluids which will be determined by the treating physician. Ultrasound measurements and other parameters listed above will be collected throughout the ED and hospital stay.
  Interventions: Device: Life Flow

INTERVENTIONS:
Device: Life Flow — LifeFlow device will be used to administer intravenous fluids in this group. LifeFlow is a FDA approved device to administer IV fluids. Subject will have a bedside ultrasound performed by the study investigator after receiving 500 ml of intravenous fluid bolus. The images will be recorded on ultrasound machine hard drive for future review. If the bedside ultrasound findings determine that the subject is not fluid responsive, subjects will be excluded from the study. If the subject is determined to be fluid responsive, the above listed outcome measures will be collected. Ultrasound will be repeated after every 500 ml bolus if the patient continues to receive IV fluids which will be determined by the treating physician. Ultrasound measurements and other parameters listed above will be collected throughout the ED and hospital stay.
  Arms: LifeFlow group

SUMMARY:
The LifeFlow rapid infusion device is a handheld manually-operated device that has been shown in early trials to increase the rate of bolus fluid infusion up to 3 times the rate of delivery attributed to conventional rapid infusion devices. The device addresses other technical barriers to fluid resuscitation, including reducing complexity and provider fatigue. LifeFlow utilizes standard IV or intraosseous (IO) vascular access devices to quickly and efficiently deliver appropriate volumes of crystalloid fluid to patients during emergent fluid resuscitation. The purpose of this study is to determine if intravenous fluids can be administered more rapidly and efficiently with the use of the LifeFlow rapid infusion device compared to the current standard techniques in adult patients who present to the Emergency Department with septic shock.

DETAILED DESCRIPTION:
Patients with conditions such as septic shock, anaphylaxis, and hypovolemic shock may require rapid fluid administration to restore blood pressure and tissue perfusion. Newly Updated Surviving Sepsis Campaign (SSC) guidelines call for patients with septic shock to receive a 30ml/kg intravenous (IV) fluid challenge within 1 hour of emergency department (ED) arrival, with improved outcomes shown with early fluid infusion. Patients with shock and severe hypotension may require even more rapid fluid treatment, up to 4ml/kg/min. While excess fluid infusion may be associated with harm, early fluid infusion for the reversal of shock can reduce the need for subsequent interventions, ultimately leading to improved patient outcomes. This may be especially true in patients with hypotension, who are at greater risk of death if not treated quickly, as a single episode of hypotension in patients with sepsis is correlated with a significantly increased risk of death.

In patients who require IV fluid bolus therapy, technical barriers such as slow infusion rates, technically complex infusion devices, and inadequate nursing resources may lead to delay in fluid administration and inadequate resuscitation. As recommended by the SSC guidelines, patients receiving fluid bolus therapy for septic shock require frequent reassessment of clinical response. With current fluid delivery techniques, the ability to reassess quickly and relate fluid administration directly to markers of hemodynamic improvement is limited.

The LifeFlow rapid infusion device is a handheld manually-operated device that has been shown in early trials to increase the rate of bolus fluid infusion up to 3 times the rate of delivery attributed to conventional rapid infusion devices. The device addresses other technical barriers to fluid resuscitation, including reducing complexity and provider fatigue. LifeFlow utilizes standard IV or intraosseous (IO) vascular access devices to quickly and efficiently deliver appropriate volumes of crystalloid fluid to patients during emergent fluid resuscitation.

The purpose of this study is to determine if intravenous fluids can be administered more rapidly and efficiently with the use of the LifeFlow rapid infusion device compared to the current standard techniques in adult patients who present to the Emergency Department with septic shock.

Primary Hypothesis

* Intravenous fluids can be administered more rapidly and efficiently with the use of the LifeFlow rapid infusion device compared to the current techniques in patients who present to the ED with hypotension and suspected septic shock Secondary Hypotheses
* Hypotensive patients receiving intravenous fluids utilizing the LifeFlow infusion device will have more rapid normalization of vital sign parameters (i.e., resolution of hypotension = MAP 65 mmHg or greater), and more rapid improvement in markers of tissue ischemia (i.e., lactate clearance) than patients receiving fluid using other techniques.
* Based on reduced ICU and hospital length of stay (LOS), the overall cost of treatment will be lower in ED patients receiving early IV fluid resuscitation with LifeFlow comparted to similar patients treated with standard techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult ED patients ≥ 18 years of age
* Patients with hypotension (Systolic Blood Pressure (SBP) < 90) mmHg or Mean Arterial Pressure (MAP) < 65 mmHg) and at least one of the following:

  * Temperature > 101 F (38.3 C) or < 96.8 F (36.0 C)
  * Respiratory Rate (RR) > 22 bpm
  * Heart Rate (HR) > 90/min
* Patients who will be determined by treating emergency physician to receive rapid fluid bolus for hypotension
* Patients with adequate cardiac windows
* EF is 35% or greater
* No increased number of B lines per rib interspace (3 or more) in multiple locations on lung ultrasound

Exclusion Criteria:

* Heart failure by history or Ejection fraction (EF) < 35 percent on pre-enrollment Point of care (POC) Echocardiogram
* History of End stage Renal disease
* History of End stage lung disease
* Lymphocyte count < 50mm/m3 or Absolute Neutrophil Count < 500
* Transferred from another facility
* Requirement for immediate surgery
* Patients with 14 Gauge catheters or larger
* Concurrently on vasopressors or inotrope therapy
* Patients or legally acceptable representatives unable to provide consent
* Non-sepsis related primary diagnosis including: acute cerebral vascular event, acute coronary syndrome, acute pulmonary edema, status asthmaticus, major cardiac arrhythmia, active gastrointestinal hemorrhage, seizure, drug overdose, burn or trauma, myocardial infarction or active hemorrhage
* Incarcerated patients
* Requirement for immediate surgery
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Time of initiation and termination of each fluid bolus administration | Up to 30 days
Volume of each fluid bolus administration | Up to 30 days

SECONDARY OUTCOMES:
Length of stay in the Emergency department, Intensive care unit, and total hospital length of stay | Up to 30 days
Resolution of abnormal blood pressure (measured at time of arrival, diagnosis and following each fluid bolus) | Up to 30 days
Assessment of Adverse effects, including rate of Intravenous fluid infiltration | Up to 30 days
Time to administration of antibiotics | Up to 30 days
Type of vasopressors used | Up to 30 days
  Epinephrine vs. Dopamine vs. Dobutamine vs. Norepinephrine
Number of subjects received a central line | Up to 30 days
Need for endotracheal intubation/mechanical ventilation | Up to 30 days
Number of ventilator-free days | Up to 30 days
Time from initial order to completion of first fluid bolus | Up to 30 days
Percent of fluid overload (FO) was calculated using the following formula: [(total fluid intake (L) - total fluid output in liters (L)) / (admission weight in kilograms)*100] | Up to 30 days
Peak Fluid overload-defined as the maximum percentage of fluid overload during the first 72 h after initiation of invasive Mechanical Ventilation | Up to 30 days
Resolution of abnormal heart rate (measured at time of arrival, diagnosis and following each fluid bolus) | Up to 30 days
Time vasopressors are started and discontinued | Up to 30 days

IPD SHARING:
Plan to Share IPD: No